CLINICAL TRIAL: NCT06730464
Title: Image-Based Prediction of Ventricular Tachycardia Events in Non-ischemic Cardiomyopathy, an International Multicenter Study - [The IMPROVE-NICM Study]
Brief Title: Image-Based Prediction of Ventricular Tachycardia Events in Non-ischemic Cardiomyopathy
Acronym: IMPROVE-NICM
Status: Recruiting | Type: Observational
Sponsor: Centro Medico Teknon (Other)
Collaborators: Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Hospital de La Luz (Other); Hospitales Universitarios Virgen del Rocio (Unknown)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Department, Centro Medico Teknon
Other Study IDs: IMPROVE-NICM
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Dilated Cardiomyopathy; Arrhythmogenic Cardiomyopathy; Ventricular Arrhythmia; Hypertrophic Cardiomyopathies
Keywords: Dilated cardiomyopathy; Non-dilated left ventricular cardiomyopathy (NDLVC); border zone channels; ventricular arrhythmias
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with non ischemic cardiomyopathies: Patients will only be recruited if they fulfill ALL the inclusion criteria:
  1. Age > 18 years.
  2. Diagnosis of non-ischemic heart disease involving the left ventricle, irrespectively of LVEF. This diagnosis includes:
     1. Dilated cardiomyopathy (DCM)
     2. Non-dilated left ventricular cardiomyopathy (NDLVC)
     3. Post-myocarditis cardiomyopathy
  3. Life expectancy of > 1 year with a good functional status.
  4. Signed informed consent.
  5. CMR already performed or scheduled for clinical purpose (standard clinical practice).
  6. No VA events at the time of the 1st LGE-CMR study.

SUMMARY:
Risk stratification for sudden cardiac death (SCD) in patients with non-ischemic cardiomyopathy (NICM) remains suboptimal. Although current guidelines rely on severe left ventricular systolic dysfunction (left ventricular ejection fraction (LVEF) < 35%) as key predictor of arrhythmic risk and clinical indication of prophylactic implantable cardioverter defibrillator (ICD), this approach seems inadequate, since registries report that only a minority of NICM ICD carriers experience an appropriate ICD shock during follow-up, whereas out-of-hospital cardiac arrests (OHCA) occur in patients with LVEF>35% in up to 80% of cases. Moreover, pivotal primary prevention trials (DANISH trial, long-term outcome of the SCD-HeFT trial) failed to demonstrate a net mortality benefit of ICD in patients with NICM.

As for most structural heart diseases (SHD), scar-related reentry has been addressed as the pathophysiological mechanism of ventricular arrhythmias (VAs) in patients with NICM, with fibrotic tissue being the substrate of this reentry. Late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) is the gold standard for the non-invasive visualization and characterization of the myocardial fibrosis and according to retrospective studies is detected in nearly 30% of patients with NICM.

In latest years, several studies and subsequent metanalyses have explored the correlation between CMR-detected LGE and occurrence of VAs, showing that presence, extent, location (septal vs lateral) and patten (focal vs multifocal vs ring-like) of non-ischemic fibrosis help in stratifying arrhythmic risk.

Nonetheless, scar heterogeneity (that is, inherent composition of dense scars vs border zone (BZ), presence of strands of viable myocardium within the scar) has been indicated as a potential novel predictor of VAs. In a recent prospective multicenter registry on patients with class I indication for cardiac resynchronization therapy (CRT) (>60% with NICM), not only scar mass, but even border zone (BZ) mass and presence of BZ channels were identified as independent predictors for VT occurrence in NICM patients.

This BZ mass and BZ channels can be automatically identified using a commercially available, post-processing imaging platform named ADAS 3D LV (ADAS3D Medical SL, Barcelona, Spain), with FDA 510(k) Clearance and CE Mark approval. Thus, CMR-derived BZ mass might be used as an automatically reproducible criterium to reclassify those patients with NICM at highest risk for developing VAs/SCD in a relatively short period of at least 2 years.

In the present cohort study, the investigators sought to: i) evaluate the usefulness of CMR-derived BZ mass measurement and identification of heterogeneous tissue channels (HTC) (among other scar characteristics derived from image post-processing) to predict the occurrence of VT events in an international, retrospective, multicenter, unselected series of patients with NICM without previous arrhythmia evidence (main study); ii) subsequently validate these predictors of VT occurrence in a prospectively-collected multicenter cohort study (substudy 1); iii) retrospectively evaluate in the subset of patients with > 1 LGE-CMR performed as part of standard clinical practice if any change in BZ mass and HTC presence occurs over time and if this correlates with occurrence of VAs (substudy 2).

DETAILED DESCRIPTION:
Primary objective To analyze the composite outcome of SCD or sustained VT (either treated by an ICD or documented by any diagnostic method) in patients with NICM and no previous arrhythmia evidence, according to their risk classification by means of number of HCT and BZ mass.

Secondary objectives Substudy 1

To validate the variables retrospectively identified to be predictors of SCD or sustained VT in a prospective cohort of consecutively enrolled patients with NICM and no previous arrhythmia evidence.

Substudy 2 To retrospectively evaluate the evolution of scar characteristics over time and their prognostic implication in the subset of patients fulfilling eligibility criteria of the main project with at least 2 LGE-CMRs available as part of their clinical follow-up.

Main study, substudy 1 and 2

To analyze the relationship between the primary outcome and other variables:

* LVEF
* Scar mass
* BZC mass
* Core mass
* Scar location
* Scar pattern
* Age
* Genotype (when this data is available)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-ischemic heart disease involving the left ventricle, irrespectively of LVEF. This diagnosis includes:

  1. Dilated cardiomyopathy (DCM)
  2. Non-dilated left ventricular cardiomyopathy (NDLVC)
  3. Post-myocarditis cardiomyopathy
* Life expectancy of > 1 year with a good functional status.
* Signed informed consent.
* At least one late gadolinium enhancement-cardiac magnetic resonance (LGE-CMR) already performed.
* No VA events at the time of the 1st LGE-CMR study.

Exclusion Criteria:

* Pregnancy.
* Life expectancy of < 1 year, or bad functional status (NYHA IV functional class).
* Other concomitant structural heart diseases (e.g. ischemic, congenital, arrhythmogenic right ventricular cardiomyopathy etc.)
* No LGE-CMR at time of enrollment or LGE-CMR data not available.
* Previously documented sustained ventricular arrhythmias at the time of 1st LGE-CMR.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dilated cardiomyopathy (DCM) or Non-dilated left ventricular cardiomyopathy (NDLVC) or Post-myocarditis cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Number of patients presenting one of sudden cardiac death, sustained ventricular arrhythmia, or defibrillator therapy. | From the inclusion date (first CMR date) up to 100 months
  The primary endpoint will be the clinical composite of sudden cardiac death, or any sustained ventricular arrhythmia, or defibrillator therapy

CONTACTS AND LOCATIONS:
Locations (4):
- Humanitas Research Hospital (Rozzano - Milan, Italy), Milan, Italy, Italy
- Hospital de la Luz, Lispon, Portugal, Portugal
- Spain (2):
  - Teknon Medical Center, Barcelona, Barcelona
  - Virgen del Rocio University Hospital, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leyva F, Taylor RJ, Foley PW, Umar F, Mulligan LJ, Patel K, Stegemann B, Haddad T, Smith RE, Prasad SK. Left ventricular midwall fibrosis as a predictor of mortality and morbidity after cardiac resynchronization therapy in patients with nonischemic cardiomyopathy. J Am Coll Cardiol. 2012 Oct 23;60(17):1659-67. doi: 10.1016/j.jacc.2012.05.054. Epub 2012 Sep 26. PMID 23021326
- [Background] Gulati A, Jabbour A, Ismail TF, Guha K, Khwaja J, Raza S, Morarji K, Brown TD, Ismail NA, Dweck MR, Di Pietro E, Roughton M, Wage R, Daryani Y, O'Hanlon R, Sheppard MN, Alpendurada F, Lyon AR, Cook SA, Cowie MR, Assomull RG, Pennell DJ, Prasad SK. Association of fibrosis with mortality and sudden cardiac death in patients with nonischemic dilated cardiomyopathy. JAMA. 2013 Mar 6;309(9):896-908. doi: 10.1001/jama.2013.1363. PMID 23462786
- [Background] Di Marco A, Brown PF, Bradley J, Nucifora G, Claver E, de Frutos F, Dallaglio PD, Comin-Colet J, Anguera I, Miller CA, Schmitt M. Improved Risk Stratification for Ventricular Arrhythmias and Sudden Death in Patients With Nonischemic Dilated Cardiomyopathy. J Am Coll Cardiol. 2021 Jun 15;77(23):2890-2905. doi: 10.1016/j.jacc.2021.04.030. PMID 34112317
- [Background] Eichhorn C, Koeckerling D, Reddy RK, Ardissino M, Rogowski M, Coles B, Hunziker L, Greulich S, Shiri I, Frey N, Eckstein J, Windecker S, Kwong RY, Siontis GCM, Grani C. Risk Stratification in Nonischemic Dilated Cardiomyopathy Using CMR Imaging: A Systematic Review and Meta-Analysis. JAMA. 2024 Sep 19;332(18):1535-50. doi: 10.1001/jama.2024.13946. Online ahead of print. PMID 39298146
- [Background] Di Marco A, Anguera I, Schmitt M, Klem I, Neilan TG, White JA, Sramko M, Masci PG, Barison A, Mckenna P, Mordi I, Haugaa KH, Leyva F, Rodriguez Capitan J, Satoh H, Nabeta T, Dallaglio PD, Campbell NG, Sabate X, Cequier A. Late Gadolinium Enhancement and the Risk for Ventricular Arrhythmias or Sudden Death in Dilated Cardiomyopathy: Systematic Review and Meta-Analysis. JACC Heart Fail. 2017 Jan;5(1):28-38. doi: 10.1016/j.jchf.2016.09.017. Epub 2016 Dec 21. PMID 28017348
- [Background] Halliday BP, Baksi AJ, Gulati A, Ali A, Newsome S, Izgi C, Arzanauskaite M, Lota A, Tayal U, Vassiliou VS, Gregson J, Alpendurada F, Frenneaux MP, Cook SA, Cleland JGF, Pennell DJ, Prasad SK. Outcome in Dilated Cardiomyopathy Related to the Extent, Location, and Pattern of Late Gadolinium Enhancement. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 2):1645-1655. doi: 10.1016/j.jcmg.2018.07.015. Epub 2018 Sep 12. PMID 30219397
- [Background] Acosta J, Fernandez-Armenta J, Borras R, Anguera I, Bisbal F, Marti-Almor J, Tolosana JM, Penela D, Andreu D, Soto-Iglesias D, Evertz R, Matiello M, Alonso C, Villuendas R, de Caralt TM, Perea RJ, Ortiz JT, Bosch X, Serra L, Planes X, Greiser A, Ekinci O, Lasalvia L, Mont L, Berruezo A. Scar Characterization to Predict Life-Threatening Arrhythmic Events and Sudden Cardiac Death in Patients With Cardiac Resynchronization Therapy: The GAUDI-CRT Study. JACC Cardiovasc Imaging. 2018 Apr;11(4):561-572. doi: 10.1016/j.jcmg.2017.04.021. Epub 2017 Aug 2. PMID 28780194
- [Background] Lehrke S, Lossnitzer D, Schob M, Steen H, Merten C, Kemmling H, Pribe R, Ehlermann P, Zugck C, Korosoglou G, Giannitsis E, Katus HA. Use of cardiovascular magnetic resonance for risk stratification in chronic heart failure: prognostic value of late gadolinium enhancement in patients with non-ischaemic dilated cardiomyopathy. Heart. 2011 May;97(9):727-32. doi: 10.1136/hrt.2010.205542. Epub 2010 Nov 20. PMID 21097819
- [Background] Halliday BP, Cleland JGF, Goldberger JJ, Prasad SK. Personalizing Risk Stratification for Sudden Death in Dilated Cardiomyopathy: The Past, Present, and Future. Circulation. 2017 Jul 11;136(2):215-231. doi: 10.1161/CIRCULATIONAHA.116.027134. PMID 28696268
- [Background] Dukkipati SR, Koruth JS, Choudry S, Miller MA, Whang W, Reddy VY. Catheter Ablation of Ventricular Tachycardia in Structural Heart Disease: Indications, Strategies, and Outcomes-Part II. J Am Coll Cardiol. 2017 Dec 12;70(23):2924-2941. doi: 10.1016/j.jacc.2017.10.030. PMID 29216988
- [Background] Poole JE, Olshansky B, Mark DB, Anderson J, Johnson G, Hellkamp AS, Davidson-Ray L, Fishbein DP, Boineau RE, Anstrom KJ, Reinhall PG, Packer DL, Lee KL, Bardy GH; SCD-HeFT Investigators. Long-Term Outcomes of Implantable Cardioverter-Defibrillator Therapy in the SCD-HeFT. J Am Coll Cardiol. 2020 Jul 28;76(4):405-415. doi: 10.1016/j.jacc.2020.05.061. PMID 32703511
- [Background] Kober L, Thune JJ, Nielsen JC, Haarbo J, Videbaek L, Korup E, Jensen G, Hildebrandt P, Steffensen FH, Bruun NE, Eiskjaer H, Brandes A, Thogersen AM, Gustafsson F, Egstrup K, Videbaek R, Hassager C, Svendsen JH, Hofsten DE, Torp-Pedersen C, Pehrson S; DANISH Investigators. Defibrillator Implantation in Patients with Nonischemic Systolic Heart Failure. N Engl J Med. 2016 Sep 29;375(13):1221-30. doi: 10.1056/NEJMoa1608029. Epub 2016 Aug 27. PMID 27571011
- [Background] Gorgels AP, Gijsbers C, de Vreede-Swagemakers J, Lousberg A, Wellens HJ. Out-of-hospital cardiac arrest--the relevance of heart failure. The Maastricht Circulatory Arrest Registry. Eur Heart J. 2003 Jul;24(13):1204-9. doi: 10.1016/s0195-668x(03)00191-x. PMID 12831814
- [Background] Kadish A, Dyer A, Daubert JP, Quigg R, Estes NA, Anderson KP, Calkins H, Hoch D, Goldberger J, Shalaby A, Sanders WE, Schaechter A, Levine JH; Defibrillators in Non-Ischemic Cardiomyopathy Treatment Evaluation (DEFINITE) Investigators. Prophylactic defibrillator implantation in patients with nonischemic dilated cardiomyopathy. N Engl J Med. 2004 May 20;350(21):2151-8. doi: 10.1056/NEJMoa033088. PMID 15152060
- [Background] Zeppenfeld K, Tfelt-Hansen J, de Riva M, Winkel BG, Behr ER, Blom NA, Charron P, Corrado D, Dagres N, de Chillou C, Eckardt L, Friede T, Haugaa KH, Hocini M, Lambiase PD, Marijon E, Merino JL, Peichl P, Priori SG, Reichlin T, Schulz-Menger J, Sticherling C, Tzeis S, Verstrael A, Volterrani M; ESC Scientific Document Group. 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2022 Oct 21;43(40):3997-4126. doi: 10.1093/eurheartj/ehac262. No abstract available. PMID 36017572